CLINICAL TRIAL: NCT00179231
Title: Olanzapine Versus Clozapine in Treatment Refractory Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 990172
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-09

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

INTERVENTIONS:
Drug: olanzapine vs. clozapine

SUMMARY:
The study involves a six-month, double-blind protocol during which eighty patients, across three sites around the country, will be randomly assigned to receive clozapine or olanzapine. The specific aims of the study are to evaluate the relative effects of olanzapine and clozapine on clinical outcomes and cognition in patients diagnosed with schizophrenia or schizoaffective disorder who have demonstrated resistance to treatment in the past.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will be males and females, ages 18-60, with a definite diagnosis by DSM-IV criteria of schizophrenia (any subtype) or schizoaffective disorder.
2. 2) All participants will be refractory according to the Kane et al (1988) criteria, with modification on the number of drug trials to at least two neuroleptic drugs at adequate doses for periods > 3 months. The criteria of Kane et al. for treatment resistance are as follows: three or more trials with antipsychotic drugs of adequate dose and duration (this is usually 4-6 weeks). The original criteria involved three types of typical neuroleptic drugs. Now, it can include any antipsychotic drug other than clozapine. Olanzapine may have been tried but the dose must not have exceeded 30 mg/day.
3. Subjects must have a PANNS-derived BPRS total score > 24 (0-6 scale) or BPRS positive subscale item score > 3 on at least two of the four items.
4. Participants will be in generally good and stable physical health.
5. Written informed consent will be obtained from all participants after a full explanation of the study and procedures. For those patients with a legal guardian, written informed consent will be obtained from the guardian, with verbal assent by the research subject.
6. Since both clozapine and olanzapine are approved agents, no specific birth control will be required for females, but advice about birth control will be provided

Exclusion Criteria:

1. Uncontrolled diabetes or hypertension.
2. Cardiac conduction abnormality or uncontrolled arrhythmia.
3. History of any blood dyscrasia, including leukemia.
4. Significant active hepatic or renal disease, including chronic hepatitis.
5. Clinically significant neurological disorder, including (but not limited to) Parkinson's disease, multiple sclerosis, seizure disorder, intracranial mass lesion (note that the presence of tardive dyskinesia is not an exclusion for participants).
6. Active cancer with or without chemotherapy within the last five years (not to include a completely excised basal cell carcinoma).
7. Active endocrinological disorder (which does not include adequately treated hypothyroidism).
8. Pregnancy or lactation.
9. An active substance use disorder within the last six months.
10. History of lack of response to an adequate trial of monotherapy with either clozapine or olanzapine in which the dose of clozapine must be > 600 mg/day or the dose of olanzapine must be > 20 mg/day; and the duration of treatment with either must be > 6 weeks.
11. History of intolerance of clozapine or olanzapine, including blood dyscrasia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80
Dates: Start 2000-05; Study Completion 2004-02

PRIMARY OUTCOMES:
There has not been an adequate of test of whether olanzapine is as effective as clozapine in treatment
resistant patients. Several recent studies suggest olanzapine may be effective in some clozapine responders as well as in treatment resistant patients. A head to head comparison is needed to clarify the relative efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Y Meltzer, M.D., Principal Investigator — Vanderbilt University Medical Center

REFERENCES:
- [Derived] Meltzer HY, Bobo WV, Roy A, Jayathilake K, Chen Y, Ertugrul A, Anil Yagcioglu AE, Small JG. A randomized, double-blind comparison of clozapine and high-dose olanzapine in treatment-resistant patients with schizophrenia. J Clin Psychiatry. 2008 Feb;69(2):274-85. doi: 10.4088/jcp.v69n0214. PMID 18232726